CLINICAL TRIAL: NCT04919928
Title: Benefits From Bimodal Fittings With Cochlear Implant and Hearing Aid vs Bilateral Hearing Aids in Patients With Asymmetric Speech Identification Scores: a Randomised Controlled Trial
Brief Title: Benefits From Bimodal Fittings With Cochlear Implant and Hearing Aid vs Bilateral Hearing Aids
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20/22868
Record Dates: First submitted 2021-05-20; First posted 2021-06-09 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Hearing Loss, Cochlear
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Cochlear Implants; Hearing Aids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bimodal solution with cochlear implant and hearing aid (CI+HA) (Experimental): This Arm will serve as the intervention group. Patients referred for evaluation of cochlear implant candidacy at Odense University Hospital will be screened for eligibility in this study and invited to participate. All patients receive new replacement HAs that can later be fitted with the CI in a bimodal solution. The patients will use the new replacement HAs for one month and are then randomized to either the intervention group with CI+HA or to the control group with continuous use of HA+HA (bilateral) for another two months. Patients randomized to the intervention group CI+HA will undergo surgery as soon as possible after randomization.
  Patients with the bimodal solution CI+HA will undergo follow-up one, three, six and twelve months after CI fitting.
  Interventions: Device: Cochlear Implant and Hearing aid in bimodal solution
- Bilateral new replacement Hearing Aids (HA+HA) (Experimental): This Arm will serve as the control group. The patients in the control group will use the new replacement HAs for one month like the intervention group and then for another three months, if they complete the study. The control group using the new replacement HAs for three months after randomization, will be offered the bimodal solution with CI to the poorer hearing ear and have the same follow-up period as the intervention group after a total of four months with new replacement HAs.
  Interventions: Device: Bilateral hearing aids

INTERVENTIONS:
Device: Cochlear Implant and Hearing aid in bimodal solution — Sixty adult participants with bilateral hearing aids (HA) referred for cochlear implantation (CI) will be included in the study. It will be patients who report limited benefit with appropriately fitted HAs in daily speech communication in quiet and in noise. The patients are depending on visual cues for successful communication.
  All the referred patients have potential optimal fitted HAs that are no longer sufficient to treat their hearing loss and to improve the daily communication. All the patients will then receive new replacement HAs with the ability to corporate with a CI for one month trial period. One month is considered as a sufficient adaptation period to new replacement HAs according to current clinical practice.
  Thirty individuals randomised to receive the intervention with CI to the poorest hearing ear.
  Arms: Bimodal solution with cochlear implant and hearing aid (CI+HA)
Device: Bilateral hearing aids — Thirty individuals randomised to the control group will continue use of the new replacement HAs another three months, thus in total of four months of use.
  Arms: Bilateral new replacement Hearing Aids (HA+HA)

SUMMARY:
Hearing-aid (HA) users with insufficient HA may be better helped with a "Bimodal solution" when replacing the HA with a Cochlear implant (CI) to the poorer hearing ear and a HA to the better hearing ear.

This randomised controlled trial can show the benefit in terms of better speech perception of the bimodal solution with CI to the poorest hearing ear compared to binaural hearing aids.

It can clarify if HAs users with insufficient HAs benefit will benefit from the bimodal solution when adding a CI to the poorer hearing ear in terms of better speech perception.

It can report the degree of perceived hearing handicap in bimodal CI-users versus bilateral HA-users by hearing -specific patient reported outcome measures (PROM) questionnaires.

And it can contribute to a specific cochlear implant candidacy criterion related to the transition from HA treatment to the CI treatment.

The purpose of this study is to determine if bimodal treatment with a hearing aid to the better hearing ear and CI to the poorer hearing ear increases the ability to understand speech and improve quality of life compared to patients that are treated with hearing aids only.

The benefit of bimodal fittings compared to the best possible bilateral HA treatment will be evaluated.

DETAILED DESCRIPTION:
Cochlear implants (CI) have been used to restore hearing in individuals with severe to profound sensorineural hearing loss. Normally, it is required that speech identification scores are below 50% in the ear considered for implantation and that the discrimination in the best-aided condition should be 60% or less. These criteria exclude many patients with asymmetrical hearing, as they have speech identification above 60% in the best-aided condition. It is necessary to investigate how patients with asymmetrical hearing can benefit from a cochlear implant in the poorer hearing ear compared to when bilaterally fitted with HAs. Furthermore, it is still unclear at which clinical relevant candidacy criterion the optimal transition from HA treatment to CI treatment in the bimodal solution occurs, as randomized studies comparing HA users and CI users do not exist. The purpose of this study is to provide clinicians with better evidence to determine if patients who benefit insufficiently from bilateral HA treatment and have a speech discrimination of the better hearing ear > 50% will benefit from a CI in the poorer hearing ear. Patients intended to include in the study will all be adults >18 years with hearing loss on both ears where cochlear implant will be considered as a treatment for the poorest hearing ear. All patients have used hearing aids on both ears for at least 1 year. The benefit of bimodal fittings compared to the best possible bilateral HA treatment is evaluated. Furthermore, it is investigated if this results in increased speech intelligibility and quality of life with a bimodal solution where a cochlear implant is used on the poorer hearing ear compared to either CI alone or bilateral hearing aids. 60 patients referred for cochlear implant at Odense University Hospital will receive new HAs that are fitted for one month. Then they will be randomized to either the intervention group with CI+HA (bimodal) or to the wait and see control group with continuous use of HA+HA (bilateral) for another three months. Participants will undergo stratified randomization depending on the hearing thresholds prior to CI surgery in the poorest hearing ear. To provide better evidence to determine if patients who benefit insufficiently from bilateral Hearing aid treatment and have a speech discrimination of the better hearing ear > 50% will benefit from a Cochlear implant in the poorer hearing ear.

Patients randomized to the intervention group CI+HA will undergo surgery as soon as possible after randomization. The control group that will use the hearing aids for an additional three months, will also be offered the bimodal solution with CI to the poorer hearing ear after total of four months with HA+HA.

Description of the cohort Inclusion criteria - Adults >18 years old. - Fluent in Danish, including reading and writing - Willing to participate in and to comply with all requirements of the protocol. - Post-lingual deafness and use one or two HAs. - Participants should have aidable hearing in the ear not considered for CI implantation - Self-reported HA use of at least eight hour per day for at least one year in both ears prior to evaluation for cochlear implantation in order to ensure, that both ears have received auditive stimulation prior to participation in the study. If possible, the validity of the self-reported hearing aid use will be checked in the HA-log by the audiology assistants. - Participants should have a PTA (0.5,1,2,4 kHz) > 40 dB HL in the ear considered for CI implantation and PTA≥40 and ≤ 70dB HL in the ear not considered for implantation. - A speech identification score

Ethics approval for the conduct of this study was obtained from the Ethics Committee Southern Denmark. 21st August 2020.

The trial will be conducted in compliance with this study protocol. All participants will undergo a process of informed consent and will be aware that participation is strictly voluntary.

Participants may withdraw from the study at any time. The project is approved by the Danish Data Protection Agency (file no. 20/22868) in Region South Denmark which is an independent authority that supervises compliance with the rules on protection of personal data. ("paraplyanmeldelse" in danish).

The study statistic analysis plan will be implemented as well.

ELIGIBILITY:
Inclusion Criteria

* Adults >18 years old.
* Fluent in Danish, including reading and writing
* Acquired post-lingual deafness
* Use of bilateral HAs for at least one year prior to evaluation for cochlear implantation candidacy. This to ensure, that both ears have received auditive stimulation
* PTA > 40 dB HL in the ear considered for CI implantation and PTA≥40 and ≤ 70dB HL in the contralateral ear in best aided condition, in quiet and in noise and in free field.
* SIS <70% in best aided condition in the ear considered for CI implantation and SIS ≥30% and ≤70% in best aided condition in the contralateral ear, in quiet and in noise and in free field.

Exclusion Criteria

* Vestibular loss in the ear not considered for CI implantation
* Surgical issues interfering with the site of implantation or anatomical contraindications such as cochlear malformations, which will be determined using MRI or CT-scans.
* Auditory nerve lesions.
* Central auditory pathway pathologies.
* Otosclerosis.
* Single sided deafness (SSD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Hearing in Noise Test (HINT) Speech identification scores | 1 hour
  Speech identification scores measured by Hearing in Noise Test (HINT). 1-100% higher is better
Speech Spatial Questionnaire (SSQ-12) | 1 hour
  Patient reported outcomes measured by Speech Spatial Questionnaire (SSQ-12). 1-10, higher is better.

SECONDARY OUTCOMES:
Dantale I | 1 hour
  Speech identification scores measured by Dantale I in quiet and noise in free field at the best aided condition. 1-100%, higher is better
Nijmegen Cochlear Implant Questionnaire (NCIQ) | 1 hour
  Patient reported outcomes measured by Nijmegen Cochlear Implant Questionnaire (NCIQ). 1-100 higher is better
Tinnitus Handicap Inventory (THI) | 1 hour
  Patient reported outcomes measured Tinnitus Handicap Inventory (THI). 1-100, lower is better
Dizziness Handicap Inventory (DHI) Patient reported outcomes measures | 1 hour
  Patient reported outcomes measured Dizziness Handicap Inventory (DHI). 1-100, lower is better.
Peak pupil dilation (PPD) | half an hour
  Peak pupil dilation measured by pupillometry and HINT, 1-100%, lower is better
Peak-time | half an hour
  Peak-time measured by pupillometry and HINT. 1-10sec, lower is better

CONTACTS AND LOCATIONS:
Overall Officials: Jesper H Schmidt, Consultant, Study Director — Ear nose and throat department/Hearing-clinic Odense University Hospital
Locations (1):
- Ear nose and throat department/Hearing-clinic Odense University Hospital, Odense, Southern Denmark, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The data sharing is described in a Data Management Plan. All Data will be anonymised.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: It is available
URL: https://dmponline.deic.dk/plans/4239

REFERENCES:
- [Derived] Jakobsen Y, Christensen Andersen LA, Schmidt JH. Study protocol for a randomised controlled trial evaluating the benefits from bimodal solution with cochlear implant and hearing aid versus bilateral hearing aids in patients with asymmetric speech identification scores. BMJ Open. 2022 Dec 29;12(12):e070296. doi: 10.1136/bmjopen-2022-070296. PMID 36581413

DOCUMENTS (2):
  • Study Protocol (2022-08-21): https://cdn.clinicaltrials.gov/large-docs/28/NCT04919928/Prot_004.pdf
  • Statistical Analysis Plan (2022-08-21): https://cdn.clinicaltrials.gov/large-docs/28/NCT04919928/SAP_005.pdf